CLINICAL TRIAL: NCT02686541
Title: Athrectomy and Drug Eluting Balloon Therapy (ADEBT) on the Femoral Popliteal Arteries
Acronym: ADEBT
Status: Approved for marketing | Type: Expanded Access
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Steven Kum Wei Cheong, Vascular Surgeon, Changi General Hospital
Other Study IDs: CG12Aug02-12
Record Dates: First submitted 2016-02-16; First posted 2016-02-19 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

INTERVENTIONS:
Device: Atherectomy followed by Drug Eluting Balloon (DEB) — Patient will undergo an intervention under anaesthesia. After pre-arthrectomy Intravascular ultrasound (IVUS) of the affected arterial segment, patient will undergo treatment with Arthrectomy, followed by post-arthrectomy IVUS analysis.
  Following arthrectomy, the affected vessel will be treated by supplementary Ranger Drug Eluting Balloon (DEB).
  During post-procedure, patients will be started on dual antiplatelets for 3 month post intervention followed by Aspirin for life unless contraindicated. Clinical follow-up, duplex ultrasound (to assess for re-stenosis) and Ankle Brachial Pressure Index (ABPI) will be performed at 1-month, 6-month and 12-month. Assessment of the symptoms, pulse, and clinical patency will be performed at each visit.

SUMMARY:
The aim of this study is to study the effects of athrectomy followed by percutaneous transluminal angioplasty using Paclitaxel coated Drug Eluting Balloon (DEB) in treating de novo or re-stenotic lesions in the femoral-popliteal artery in patients with symptomatic peripheral vascular disease in an Asian population. The intention is to study the effects of debulking athrectomy followed by application of DEBs to prevent restenosis, resulting in improved patency rates The study will prospectively recruit 8 cases treated with athrectomy followed by DEB. This project is a pilot to investigate the effects of athrectomy and DEB in reducing re-stenosis rates. It will be a primer for a larger scale randomized controlled trial (RCT) involving multiple institutions to demonstrate the benefit of athrectomy and DEB technology to treat de novo versus plain balloon angioplasty with bail-out stenting, which is currently the most commonly used modality to treat femoral-popliteal lesions. There are no studies combining the effect of rotational athrectomy and DEBs.

DETAILED DESCRIPTION:
Patient will undergo an intervention under anaesthesia. After common femoral artery sheath access, a diagnostic angiogram will be performed. After pre-arthrectomy Intravascular ultrasound (IVUS) of the affected arterial segment, patient will undergo treatment of the lesion with arthrectomy, followed by post-arthrectomy IVUS analysis. Following arthrectomy, the affected vessel will be treated by supplementary Ranger Drug Eluting Balloon (DEB). During post-procedure, patients will be started on dual antiplatelets for 3 months followed by Aspirin for life unless contraindicated. Clinical follow-up, duplex ultrasound (to assess for re-stenosis) and Ankle Brachial Pressure Index (ABPI) will be performed at 1-month, 6-month and 12-month post intervention. Assessment of the symptoms, pulse, and clinical patency will be performed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ≥ 50% stenosis or occlusions of the femoral or popliteal artery (including below knee popliteal artery) proven on 2 views during angiography of Rutherford stage 2-6 lesions
* At least one tibial vessel runoff
* Life expectancy >1 year

Exclusion Criteria:

* Subintimal recanalisation of the affected de novo artery which would preclude treatment with athrectomy
* Patient unwilling or unlikely to comply with follow-up schedule
* GFR <30 ml/min
* Planned major index limb amputation
* Acute limb ischaemia
* Untreated ipsilateral iliac artery stenosis ≥ 50
* Previous atherectomy, brachytherapy or cryoplasty of the affected arterial segment
* Severe flow limiting dissection or residual stenosis >50% post initial athrectomy requiring supplementary stenting
* Female patients of childbearing potential

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2015-04; Primary Completion 2017-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kum, MBBS, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore